CLINICAL TRIAL: NCT05634707
Title: A Randomized Surgical Window of Opportunity Study With Dose Escalation to Evaluate Whether Oral Fluoxetine Can Induce Cytotoxic Lysosomal Stress and Enhance Temozolomide Efficacy in Clinical Glioma
Brief Title: Evaluation of Fluoxetine and Cytotoxic Lysosomal Stress in Glioma (FLIRT)
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00110628
Record Dates: First submitted 2022-11-22; First posted 2022-12-02 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Primary Brain Tumor; Brain Tumor, Recurrent
Keywords: Brain tumor; Fluoxetine; Prozac; Recurrent; Glioma; Temozolomide; Tumor resection; Tumor biopsy; Mustafa Khasraw; Pro00110628
MeSH Terms: conditions — Brain Neoplasms; Recurrence; Glioma | interventions — Fluoxetine; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluoxetine pre-surgery (Experimental): Patients randomized to the experimental arm will receive fluoxetine at 20 mg/day for 5 days (initiation dose) followed by a maintenance dose of 40 mg/day starting on Day 6 (dose level 1) or 60 mg/day starting on Day 6 (dose level 2).
  Interventions: Drug: Fluoxetine
- Temozolomide pre-surgery (Active Comparator): Temozolomide pre-surgery (control) arm will receive 50 mg/m2 temozolomide daily for 7 days (Days 1-7), followed by resection or biopsy 21 days after initiation of the temozolomide cycle.
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Fluoxetine — Patients randomized to the experimental arm will receive fluoxetine 20mg/day for 5 days before escalation to a maintenance dose at day 6. On day 6, patients will start treatment with 50 mg/m2 TMZ daily for 7 days (Days 6-12)
  * Arm 2A (n=10) - Escalate to maintenance 40mg/day fluoxetine on day 6
  * Arm 2B (n=10) - This arm will be opened as long as there are less than 3/10 dose limiting toxicities in Arm 2A. Patients will escalate to maintenance 60mg/day fluoxetine on day 6
  Arms: Fluoxetine pre-surgery
Drug: Temozolomide — Patients randomized to the control arm will receive 50 mg/m2 temozolomide daily for 7 days (Days 1-7), followed by resection or biopsy 21 days after initiation of the temozolomide cycle.
  Arms: Temozolomide pre-surgery

SUMMARY:
The purpose of this research study is to determine if fluoxetine increases lysosomal stress in patients with recurrent IDHwt glioma by evaluating LAMP1 expression in tumor samples obtained pre-resection via biopsy and during surgery. Lysosomes are organelles (structures in cells) that contain digestive enzymes (substances that break down chemicals) that help keep the cells free of extra or worn out cell parts. Fluoxetine, a drug approved by the FDA to treat problems like depression and anxiety, can cause changes to structures in cells called lysosomes that then improve how well the chemotherapy drug temozolomide (TMZ) kills cancer cells in the brain.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether oral fluoxetine can induce lysosomal stress and enhance Temozolomide (TMZ)-induced cell death in patients diagnosed with recurrent malignant glioma. The primary objective is to determine if fluoxetine increases lysosomal stress in patients with recurrent IDHwt glioma by evaluating LAMP1 expression in tumor samples obtained pre-resection via biopsy and during surgery. Following consent, an optional biopsy may be performed to confirm recurrence of high-grade glioma. Recurrent glioma patients for whom retreatment with TMZ is appropriate and who are able to undergo tumor resection after 1 cycle of temozolomide will be enrolled in this study. Following enrollment, patients will randomly be assigned to (1:2) a study arm: control (n=10) or experimental (n=20). Within the experimental arm, two maintenance dose levels of fluoxetine are planned - 40mg OD (n=10) and 60mg OD (n=10). Patients randomized to the control arm will receive only 50 mg/m2 TMZ daily for 7 days (Days 6-12), followed by resection 21 days after initiation of the TMZ cycle. Patients randomized to the experimental arm will receive fluoxetine at 20 mg/day for 5 days (loading initiation dose) followed by a maintenance dose of 40 mg/day starting on Day 6 (dose level 1) or 60 mg/day starting on Day 6 (dose level 2) This truncated initiation period of fluoxetine has been discussed with the psychiatry department at Duke University Hospital and has been judged to be safe given the additional monitoring precautions that are being included as part of this study. On Day 6, patients will start treatment with 50 mg/m2 TMZ daily for 7 days (Days 6-12). Resection will occur 21 days after initiation of the TMZ cycle on Day 27. Patients will remain on their assigned dose of fluoxetine through resection and follow-up, as long as the treatment regimen is tolerated. The change between baseline and post-resection will be computed to determine if co-administration of fluoxetine and TMZ will result in increased expression of LAMP1 on resected glioma cells. Within each group, a Wilcoxon signed-rank test will be conducted to determine if there are significant within group changes. A Kruskal-Wallis test will compare the three patient groups (Control Group, Fluoxetine Group [low-dose], Fluoxetine Group [high-dose]) with respect to these changes. If data suggests that parametric method are appropriate, then analysis of variance and a paired t-test will be conducted. Risks commonly associated with fluoxetine include nausea, diarrhea, lack of appetite, dry mouth, upset stomach or heartburn, constipation, insomnia, anxiety, nervousness, drowsiness, tremor, unusual dreams, headaches, dizziness, yawning, swelling of face, low body temperature, sexual dysfunction, rash, hives and itching, sweating, flu-like symptoms, sore throat, stuffy nose, and fever.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 24 years of age Note: Fluoxetine has a warning about suicidal thoughts in children, adolescents, and young adults. Short-term studies did not show an increase in the risk of suicidality with antidepressants compared to placebo in adults beyond age 24.
2. Patients with recurrent glioma
3. Tumor volume ≥ 1 cm3
4. Clinical indication for craniotomy for biopsy and resection of the lesion
5. Clinical indication for repeat treatment with Temozolomide
6. Karnofsky Performance Status (KPS) > 70%
7. Adequate organ function: platelets > 100,000/µL, hemoglobin >9 gm/dL, ANC > 1000/µL; creatinine < 1.5x upper limit of normal (ULN), total bilirubin < 1.5x ULN, AST/ALT < 2.5x ULN within 72 hours prior to first administration of Fluoxetine
8. Able to undergo MRI brain with and without contrast
9. If the patient is a sexually active female of childbearing potential, whose partner is male, or if the patient is a sexually active male, whose partner is a female of childbearing potential, the patient must use appropriate contraceptive measures for the duration of the treatment and for 6 months afterwards. Female patients of childbearing potential must have a negative serum pregnancy test at the time of screening and within 48 hours of starting the infusion of the study drug.
10. Signed informed consent approved by the Institutional Review Board

Exclusion Criteria:

1. Patients currently taking or who have taken any other anti-depressant medication within the past year
2. Patients currently taking psychotropic agents or who have taken other psychotropic agents within the past 7 days
3. Patients with any history of mood/psychotic/substance use disorders
4. Prior, unrelated malignancy requiring current active treatment except for cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin
5. Patients who are pregnant or breastfeeding
6. Patients with contrast-enhancing tumor crossing the midline, multifocal tumor, infratentorial tumor, tumor in eloquent brain regions, extensive tumor dissemination (subependymal or leptomeningeal), or in unsafe brain regions per the opinion of the treating neurosurgeon
7. Patients with worsening neurologic deficits, clinically significant increased intracranial pressure (e.g., impending herniation), uncontrolled seizures, or requirement for immediate palliative treatment
8. Unstable systemic disease in the opinion of the treating physician
9. Less than 12 weeks from radiation therapy, unless progressive disease outside of the radiation field or 2 progressive scans at least 4 weeks apart or histopathologic confirmation of recurrent tumor
10. Treated with immunotherapeutic agents within 4 weeks, alkylating agents within 4 weeks, nitrosoureas within 6 weeks, or non-alkylating chemotherapy within 2 weeks before enrollment, unless the patient has recovered from the expected toxic effects of such therapy
11. Treated with antiangiogenic agents (i.e., bevacizumab) within 4 weeks before biopsy
12. Patients who have developed disease progression while receiving temozolomide treatment are not eligible
13. Patients with allergy to fluoxetine
14. Patients with known cardiac disease, predisposing to long QT syndrome
15. Patients with diabetes mellitus, epilepsy, history of bleeding disorders, history of mania or susceptibility to angle-closure glaucoma
16. Patients with a history or who develop significant hyponatremia (serum sodium less than 130mmol/L)
17. Patients with a history of bipolar disorder or schizoaffective disorder
18. Patients with a history of seizure disorder prior to onset of their primary glioma
19. Patients who are currently taking or have taken in the past 2 months: Monoamine Oxidase Inhibitors (MAOI), Pimozide, Thioridazine, Drugs metabolized by the CYP2D6 pathway, Tricyclic Antidepressants, Antipsychotics, Serotonergic Drugs, Triptans, Tryptophan, Anticoagulant drugs (e.g., NSAIDs, aspirin, warfarin), Olanzapine
20. Patients who demonstrated thrombocytopenia following prior treatment with TMZ (platelets < 50,000/µL)

Min Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-08-05 (Actual); Primary Completion 2026-12-05 (Estimated); Study Completion 2027-06-05 (Estimated)

PRIMARY OUTCOMES:
Change in LAMP1 expression in tumor samples obtained pre-resection via biopsy and during surgery | baseline, 1 month
  Determine if fluoxetine increases lysosomal stress in patients with recurrent IDHwt glioma by evaluating LAMP1 expression in tumor samples obtained during surgery or biopsy

SECONDARY OUTCOMES:
Proportion of patients with partial or complete response at the time of surgical resection | 1 month
  Estimate the objective radiographic response rate
Serum levels of fluoxetine using LC-MS/MS quantification | 1 month
  Compare groups (Control Group, Fluoxetine Group (low-dose), Fluoxetine Group (high-dose)) with respect to serum levels of fluoxetine.
Serum levels of norfluoxetine using LC-MS/MS quantification | 1 month
  Compare groups (Control Group, Fluoxetine Group (low-dose), Fluoxetine Group (high-dose)) with respect to serum levels of norfluoxetine.
Intra-tumoral levels of fluoxetine using LC-MS/MS quantification | 1 month
  Compare groups (Control Group, Fluoxetine Group (low-dose), Fluoxetine Group (high-dose)) with respect to intra-tumoral levels of fluoxetine.
Intra-tumoral levels of norfluoxetine using LC-MS/MS quantification | 1 month
  Compare groups (Control Group, Fluoxetine Group (low-dose), Fluoxetine Group (high-dose)) with respect to intra-tumoral levels of norfluoxetine.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Khasraw, MBChB, MD, FRCP, FRACP, Principal Investigator — Duke University
Locations (4):
- United States (4):
  - UC San Diego Moores Cancer Center, San Diego, California
  - Stanford Cancer Institute, Stanford, California
  - NYU Langone Health, New York, New York
  - The Preston Robert Tisch Brain Tumor Center at Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Preston Robert Tisch Brain Center at Duke University — https://tischbraintumorcenter.duke.edu/
- See also: Duke Health — http://www.dukehealth.org/clinical-trials